CLINICAL TRIAL: NCT07022015
Title: Predictive Risk Factors for Postoperative Pancreatic Fistula After Pancreaticoduodenectomy for Malignancy.
Brief Title: Predictive Risk Factors for Pancreatic Fistula After Pancreaticoduodenectomy
Acronym: POPF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Minia University (Other)
Responsible Party: Principal Investigator, Saleh Khairy Saleh MD, Lecturer, Minia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1438/2025
Record Dates: First submitted 2025-06-05; First posted 2025-06-15 (Actual); Last update posted 2025-06-22 (Actual); Status verified 2025-06

CONDITIONS: Pancreas Cancer; Pancreas Neoplasm; Pancreatic Fistula; Pancreas Adenocarcinoma; Periampullary Cancer; Periampullary Carcinoma; Resectable Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Clinically relevant postoperative pancreatic fistula (Other): patients who developed clinically relevant postoperative pancreatic fistula after pancreaticoduodenectomy
  Interventions: Procedure: pancreaticoduodenectomy procedure

INTERVENTIONS:
Procedure: pancreaticoduodenectomy procedure — Pancreaticoduodenectomy operation
  Other Names: PD

SUMMARY:
Pancreaticoduodenectomy (PD) is a complex procedure performed in patients with malignant or benign tumors of the pancreatic head and periampullary region, associated with high morbidity and mortality. Postoperative pancreatic fistula (POPF) is the most common and clinically significant complication following PD. In this study, the investigators aim to determine the predictive risk factors for clinically related postoperative pancreatic fistula (CR-POPF) in the preoperative, intraoperative and postoperative period in patients that underwent PD. The total number of 100 participants expected to be included in this research who underwent PD between 2025 and 2026.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy (PD) is a complex procedure performed in patients with malignant or benign tumors of the pancreatic head and periampullary region, associated with high morbidity and mortality rates. Despite dramatic advancements in surgical techniques and perioperative management, reported morbidity and mortality rates following PD are 41.56% and 2.88%, respectively, which remain unsatisfactory. Postoperative pancreatic fistula (POPF) is the most common and clinically significant complication following PD. Therefore, accurate and timely prediction of POPF after PD is necessary to reduce secondary mortality from serious complications and optimize individual patient treatment decisions. This study aimed to determine the predictive risk factors for clinically related postoperative pancreatic fistula (CR-POPF) in the preoperative, intraoperative and postoperative period in patients that underwent PD.

ELIGIBILITY:
Inclusion Criteria:

* Patients with resectable distal common bile duct carcinoma, periampullary carcinoma, duodenal carcinoma, and carcinoma of the head of the pancreas.
* Patients meeting the curative treatment intent in accordance with clinical guidelines:

  * No evidence of metastasis.
  * Radiological non-involvement of superior mesenteric vein & portal vein.
* American Society of Anesthesiologists (ASA) scores I & II.
* Patients aged > 18 years.
* Ability to understand and the willingness to sign a written informed consent document
* Agreement to complete the study

Exclusion Criteria:

* Unfit patients for surgery due to severe medical illness.
* Inoperable patients with distant metastases, including peritoneal, liver, distant lymph node metastases, and involvement of other organs.
* Irresectable tumors in diagnostic laparoscopy.
* History of other malignant disease.
* Pregnant or breast-feeding women.
* Patients with serious mental disorders.
* Patients with vascular invasion and requiring vascular resection as evaluated by the multidisciplinary team according to abdominal imaging data.
* Pancreatoduodenectomy for other diagnosis like cystic lesions, benign tumors or chronic calcific pancreatitis
* Patients refused to participate in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-06-20 (Actual); Primary Completion 2026-06-20 (Estimated); Study Completion 2026-07-20 (Estimated)

PRIMARY OUTCOMES:
Incidence of clinically relevant post operative pancreatic fistula | 10 days
  A drainage fluid of any measurable volume with an amylase level more than three times the upper normal serum level on or after the 3rd postoperative day

CONTACTS AND LOCATIONS:
Overall Officials: Saleh K Saleh, MD, Principal Investigator — Minia University
Locations (1):
- Liver and GIT hospital , Minia University, Minya, Minya Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No